CLINICAL TRIAL: NCT03939403
Title: Conventional Ovarian Stimulation vs. Single Injection Stimulation of Corifollitropin Alfa in Oocyte Donor. A Randomized Clinical Trial. TAIL Study
Brief Title: Conventional Ovarian Stimulation vs. Single Injection Stimulation of Corifollitropin Alfa in Oocyte Donor
Acronym: TAIL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto Bernabeu (Other)
Responsible Party: Principal Investigator, Joaquín Llácer, Principal Investigator, Instituto Bernabeu
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IB-0319-002
Record Dates: First submitted 2019-05-03; First posted 2019-05-06 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Ovarian Stimulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 7-days pill free interval (Experimental)
  Interventions: Drug: Time of administration of Corifollitropin Alfa
- 5-days pill free interval (No Intervention)

INTERVENTIONS:
Drug: Time of administration of Corifollitropin Alfa — The used treatment will be identical in both arms. The difference between the groups will be the moment of beginning of the stimulation as well as the later administration of more FSH activity.
  The control grup will receive the treatment on the 5th day after the cessation of hormonal contraceptive use. The used treatment will be identical in both arms. The difference between the groups will be the moment of beginning of the stimulation as well as the later administration of more FSH activity.
  The intervention grup will receive the treatment on the 7th day after the cessation of hormonal contraceptive use.
  Arms: 7-days pill free interval

SUMMARY:
This study aims to study the efficiency of using a single injection of Corifollitropin alfa for ovarian stimulation by initiating administration late and without further administration of follicle-stimulating hormone after the 7th day of stimulation compared to conventional ovarian stimulation using Corifollitropin alfa (drug administration 5 days after cessation of hormonal contraceptive and supplementation with follicle-stimulating hormone daily administration from the 8th day of stimulation).

This a controlled randomized clinical study and 180 patients will be recruited (90 per arm) and the primary study outcome is the number of obtained oocytes.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for oocyte donation program
* Age between 18 and 32 years old
* BMI >18 and <30
* Antral follicle count >12 (summing both ovaries)
* Presence of both ovaries
* Ability to participate in and comply with study protocol
* Signed informed consent
* No treatment with ovulation stimulators in the 3 months prior to the start of stimulation.

Exclusion Criteria:

* Diagnosis of endometriosis at any stage
* AFC >20
* Polycystic ovary syndrome
* Concurrent participation in another study

Ages: 18 Years to 32 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2019-11-18 (Actual); Primary Completion 2021-05-08 (Actual); Study Completion 2021-05-08 (Actual)

PRIMARY OUTCOMES:
Number of oocytes | At the end of stimulation
  Number of oocytes after stimulation

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Bernabeu, Alicante, Spain

IPD SHARING:
Plan to Share IPD: Undecided